CLINICAL TRIAL: NCT07253974
Title: Prospective Evaluation of Atrial Fibrillation-Related Stroke Patients in Rehabilitation Program (PEARL), an Observational Cohort Study. TARGET: Health Virtual Twins for the Personalised Management of Stroke Related to Atrial Fibrillation".
Brief Title: Prospective Evaluation of Atrial Fibrillation-Related Stroke Patients in Rehabilitation Program (PEARL), an Observational Cohort Study
Acronym: PEARL
Status: Recruiting | Type: Observational
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/11172/I_PEARL; n.101136244 (Other Grant/Funding Number: European Union's Horizon Europe)
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: STROKE; Rehabilitation Outcome; Brain Disease; Cardiovascular Disease Acute; Hemiplegia and/or Hemiparesis Following Stroke; Disability Physical
Keywords: functional outcomes; stroke; disability; rehabilitation; high intensity rehabilitation program
MeSH Terms: conditions — Stroke; Brain Diseases | interventions — Occupational Therapy; Deglutition; Language Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High Intensity Rehabilitation program: NIHSS 3-13, MRS historic ( pre-Stroke)1-2, Cognitive status : preserved
  Interventions: Other: Rehabilitation program based on Physiotherapy, occupational therapy and swallow and language therapy
- Moderate Intensity Rehabilitation program: NIHSS >13 or MRS historic ( pre-Stroke)<3
  Interventions: Other: Rehabilitation program based on Physiotherapy, occupational therapy and swallow and language therapy

INTERVENTIONS:
Other: Rehabilitation program based on Physiotherapy, occupational therapy and swallow and language therapy — Rehabilitation will begin in the acute care setting. After discharge from the stroke unit, all patients needing inpatient rehabilitation will undergo standard therapies (physiotherapy, occupational therapy, speech therapy, social work and neuropsychology) in an Intensive Inpatient Rehabilitation Facilities (IRF) or a Skilled Nursing Facilities (SNF). The choice of setting will depend on age, functional level before stroke, stroke impairment severity and cognitive and medical status. In the High-Intensity Rehabilitation program in IRF, patients will undergo at least 3 sessions of Inpatient Physiotherapy (PT), Occupational Therapy (OT) and Speech-Language Pathologist (SLT). In the moderate-intensity rehabilitation program delivered in SNFs, patients will receive approximately one or two session of therapy per day, including PT, OT, and SLT, when indicated.

SUMMARY:
The goal of this observational study is to determine if rehabilitation program intensity impacts functional recovery and specific needs in adult ischemic stroke patients who require inpatient rehabilitation. The main questions it aims to answer are:

Do patients with stroke of Atrial-related subtypes (AFRS) have distinct rehabilitation needs and functional outcomes compared to non-AFRS patients? Does higher-intensity inpatient rehabilitation (3-5 sessions/day) result in better functional recovery at six months (measured by the Barthel Index) than moderate-intensity programs (1 session/day)? The study is non-invasive, does not interfere with usual care. The investigators' ultimate goal is to enhance the understanding of recovery after following different rehabilitation usual programs.

DETAILED DESCRIPTION:
Introduction: Rehabilitation is recognised as a cornerstone of the recovery stroke care period. The intensity of therapy is related to functional recovery. Longitudinal studies investigating differences in short- and long-term outcomes of ischemic and hemorrhagic strokes are scarce. The investigators do not know whether AFRS have specific rehabilitation needs or different functional outcomes from non-AFRS. Identifying differences in aetiology and stroke recovery can help the scientific community to develop predictive models of recovery optimizing available resources.

Methods and analysis: In this prospective observational study stroke patients will be recruited in the Stroke Unit of one tertiary hospital. Patients discharged from the Stroke Unit who need inpatient rehabilitation will be allocated to two rehabilitation centers with programs of different intensity: High-intensity (3-5 session daily) or Moderate-intensity (1session daily) based on Rehabilitation Catalan Stroke Rehabilitation Plan.

Screening criteria are based on Current clinical items: age, prior functional level, neurological impairment and cognitive and medical status.

After discharge from the stroke unit, the post-acute inpatient care services for stroke patients include rehabilitation facilities and long-term care hospitals. Intensive inpatient programs provide hospital-level care and offer rehabilitation (RHB) at least 3 sessions of therapy per day 6 days a week, aiming at regaining lost body functions and recovering autonomy in basic activities of daily life. Patients treated in these inpatient rehabilitation facilities have better functional outcomes and higher rates of return to community living than those treated in general wards or long-term care hospitals. Long-term care centres and Nursing Facilities offer Moderate-intensity programs, which consist of 1 session of rehabilitation daily.

In patients with moderate-to-severe post-stroke acute deficits, there is high inter-individual variability in recovery which makes predicting outcomes much more difficult. Accumulated evidence suggests that both initial motor impairment and long-term motor outcome depend on the severity of corticospinal tract (CST) damage and the integrity of alternative motor fibres. Measurements extracted from magnetic resonance imaging (MRI), diffusion tensor (DTI), and functional imaging (fMRI) provide comprehensive in vivo metrics of local microstructural and functional connectivity properties of brain tissue. Despite these advances, in clinical practice, there is no validated gold standard for predicting functional outcomes after stroke. Nevertheless, to date 21 stroke registries across 19 different countries have been documented; and some clinical trials aimed at developing data-driven prediction models are currently underway, These efforts reflect a growing interest among RHB- teams in optimizing interventions throughout the stroke care continuum.

Differences between aetiology Typically published studies do not differentiate between stroke aetiology, at most they may define ischaemic or haemorrhagic events. Longitudinal studies investigating differences in short- and long-term outcomes of strokes according to their aetiology are scarce. Atrial fibrillation (AF) affects approximately 1-2% of the general population and is associated with a 5-fold increased risk of stroke.

In the Nationwide Danish Stroke Registry analysing 14.662 patients with atrial fibrillation related stroke (AFRS) experienced more severe strokes and higher morbidity and mortality rates, with a final greater disability at discharge. However, the investigators do not have information on the rehabilitation needs and final functional results in specific AFRS, but some recent studies suggests that AF type and related cardiac markers could serve as predictors for poor functional and cognitive outcomes. Identifying differences in aetiology and stroke recovery can help the scientific community to develop predictive models of recovery optimizing available resources.

The PEARL study is part of the TARGET project, a Horizon Europe funded programme which includes risk prediction, diagnosis and management of AF-related stroke (https://target-horizon.eu/). One of the aims of the project focuses on identifying predictors of functional independence and quality of life in AFRS survivors and facilitating personalisation of rehabilitation.

The PEARL study, as part of the TARGET project, is a prospective observational cohort study conducted over a two-year period in a tertiary Rehabilitation department. The study aims to collect data on the recovery trajectory of patients with acute stroke, with a particular focus on comparing individuals with atrial fibrillation-related stroke (AFRS) to those without, in terms of functional outcomes following admission to either high- or moderate-intensity rehabilitation programmes.

Ethics and dissemination: National and international research ethics guidelines will be followed, including the Deontological Code of Ethics, Declaration of Helsinki, and Spain's confidentiality law concerning personal data (Ley Orgánica 15/1999, 13 December, Protección de Datos de Carácter Personal). The study has received approval by the local Ethics Committee (N. 2023/11172/I) and participants will give written consent prior to study inclusion.It has been registered on clinicaltrials.gov

ELIGIBILITY:
Inclusion Criteria:> 18 a, first-ever intracerebral ischemic stroke

-

Exclusion Criteria:

* intracranial haemorrhage, symptomatic hemorrhagic transformation, new infarcts after the initial stroke or other neurological or psychiatric conditions.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ischemic stroke patients admitted to the Stroke Unit
Sampling Method: Non-Probability Sample
Enrollment: 213 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2026-11-11 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Barthel improvement | The assessment will be performed at inpatient rehabilitation at Baseline, at admission to the rehabilitation dept (T0), at 1-month follow-up (T1-discharge), and at 3-month (T2) and 6-month (T3) follow-ups after the acute event.
  To compare 6-month functional outcomes (Barthel Index) between AFRS and non-AFRS patients within high-intensity and moderate-intensity rehabilitation programs.
  Unit of Measure: Score (0-100)

SECONDARY OUTCOMES:
Functional outcomes pre and after rehabilitation program | From enrollment to 6-month follow-up.
  To evaluate differences in occupational therapy, physiotherapy, speech therapy, and cognitive outcomes between AFRS and non-AFRS patients:
Change Barthel from Baseline to 6-month follow-up outcomes | From enrollment to 6-month after stroke event
  To compare 6-month functional outcomes (Barthel Index) between AFRS and non-AFRS patients within high-intensity and moderate-intensity rehabilitation programs.
Functional Ambulation Category (FAC) | Baseline (T0), 1-mo follow-up (discharge--T1) and follow-up at 3-month (T2) and six-month (T3) after the acute event
  Ambulation ability classification. Ordinal category (0-5)
Trunk Control Test (TCT) | Baseline (T0), 1-mo follow-up (discharge--T1) and follow-up at 3-month (T2) and six-month (T3) after the acute event
  Assesses trunk control in stroke patients Score (0-100)
Berg Balance Scale (BBS) | Baseline (T0), 1-mo follow-up (discharge--T1) and follow-up at 3-month (T2) and six-month (T3) after the acute event
  Assessment of static and dynamic balance. Score (0-56)
Timed Up and Go (TUG) | Baseline (T0), 1-mo follow-up (discharge--T1) and follow-up at 3-month (T2) and six-month (T3) after the acute event
  Functional mobility test: sit-to-stand, ambulation, turning, and return Unit of Measure: Seconds
Gait Velocity (10-Meter Walk Test) | Baseline (T0), 1-mo follow-up (discharge--T1) and follow-up at 3-month (T2) and six-month (T3) after the acute event
  Walking speed over 10 meters. Unit of Measure: Meters/second (m/s)
9-Hole Peg Test (9HPT) | Baseline (T0), 1-mo follow-up (discharge--T1) and follow-up at 3-month (T2) and six-month (T3) after the acute event
  Fine motor dexterity test Unit of Measure: Seconds
Handgrip Strength | Baseline (T0), 1-mo follow-up (discharge--T1) and follow-up at 3-month (T2) and six-month (T3) after the acute event
  Upper-limb strength measured via dynamometry. Unit of Measure: Kilograms (kg)
Montreal Cognitive Assessment (MoCA) | Baseline (T0), follow-up at 3-month (T2) and six-month (T3) after the acute event
  Cognitive screening for multiple domains. Unit of Measure: Score (0-30)
EQ-5D-5L | Baseline (T0), six-month (T3) after the acute event
  Quality-of-life measure including index score and VAS Unit of Measure: Index score and VAS (0-100)
Dysphagia Assessment (Volume-Viscosity Swallow Test) | Baseline (T0)
  Evaluation of swallowing safety and efficacy. Unit of Measure: Categorical (normal / impaired)
Aphasia Presence | Baseline (T0)and six-month (T3) after the acute event
  Aphasia recorded by speech-language pathology. Unit of Measure: Dichotomous (yes/no)
NIH Stroke Scale (NIHSS) | Baseline (T0)
  Quantifies neurological deficit in acute stroke. Unit of Measure: Score (0-42)
Modified Rankin Scale (mRS) | Baseline (T0), 1-mo follow-up (discharge--T1) and follow-up at 3-month (T2) and six-month (T3) after the acute event
  Global disability scale Unit of Measure: Score (0-6)
Hospital Anxiety and Depression Scale (HADS) | Baseline (T0), and follow-up at six months (T3) after the acute event
  Measures symptoms of anxiety and depression. Unit of Measure: Score (0-21 for anxiety; 0-21 for depression)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Guillen-Sola, MD, PHd, Principal Investigator — Research Rehabilitation Group, IMIM
Locations (1):
- Rehabilitation Research Group, IMIM, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
This study is part of the EU Horizon 2020 TARGET project, following its DMP to ensure data is handled ethically, legally, and sustainably in line with FAIR principles (Findability, Accessibility, Interoperability, Reusability). The plan ensures systematic organization, quality consistency via standardized procedures, and compliance with GDPR, national laws, and EU requirements. Personal data is processed securely, only when necessary for project objectives, with approvals and written consent from participants. Methods include interviews, surveys, workshops, and questionnaires. Data is stored with robust backup and preservation strategies to prevent loss and ensure future usability. Sharing is (currently) restricted to the consortium under a signed data transfer agreement, with external sharing undecided. Data not publicly available includes: third-party data without permission for public release, data compromising IP protection, and participant data that cannot be fully anonymized.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: November 2024-December 2027

REFERENCES:
- [Background] Tracz J, Gorczyca-Glowacka I, Rosolowska A, Wozakowska-Kaplon B. Long-Term Outcomes after Stroke in Patients with Atrial Fibrillation: A Single Center Study. Int J Environ Res Public Health. 2023 Feb 16;20(4):3491. doi: 10.3390/ijerph20043491. PMID 36834183
- [Result] Alcusky M, Ulbricht CM, Lapane KL. Postacute Care Setting, Facility Characteristics, and Poststroke Outcomes: A Systematic Review. Arch Phys Med Rehabil. 2018 Jun;99(6):1124-1140.e9. doi: 10.1016/j.apmr.2017.09.005. Epub 2017 Sep 28. PMID 28965738
- [Result] Shah S, Vanclay F, Cooper B. Improving the sensitivity of the Barthel Index for stroke rehabilitation. J Clin Epidemiol. 1989;42(8):703-9. doi: 10.1016/0895-4356(89)90065-6. PMID 2760661
- [Result] Ortega-Martorell S, Olier I, Ohlsson M, Lip GYH; TARGET Consortium. TARGET: A Major European Project Aiming to Advance the Personalised Management of Atrial Fibrillation-Related Stroke via the Development of Health Virtual Twins Technology and Artificial Intelligence. Thromb Haemost. 2025 Jan;125(1):7-11. doi: 10.1055/a-2438-5671. Epub 2024 Oct 14. No abstract available. PMID 39401519
- [Result] Vinding NE, Kristensen SL, Rorth R, Butt JH, Ostergaard L, Olesen JB, Torp-Pedersen C, Gislason GH, Kober L, Kruuse C, Johnsen SP, Fosbol EL. Ischemic Stroke Severity and Mortality in Patients With and Without Atrial Fibrillation. J Am Heart Assoc. 2022 Feb 15;11(4):e022638. doi: 10.1161/JAHA.121.022638. Epub 2022 Feb 12. PMID 35156393
- [Result] Stinear CM, Ward NS. How useful is imaging in predicting outcomes in stroke rehabilitation? Int J Stroke. 2013 Jan;8(1):33-7. doi: 10.1111/j.1747-4949.2012.00970.x. PMID 23280267
- [Result] Deutsch A, Granger CV, Heinemann AW, Fiedler RC, DeJong G, Kane RL, Ottenbacher KJ, Naughton JP, Trevisan M. Poststroke rehabilitation: outcomes and reimbursement of inpatient rehabilitation facilities and subacute rehabilitation programs. Stroke. 2006 Jun;37(6):1477-82. doi: 10.1161/01.STR.0000221172.99375.5a. Epub 2006 Apr 20. PMID 16627797
- [Result] Wang H, Camicia M, DiVita M, Mix J, Niewczyk P. Early inpatient rehabilitation admission and stroke patient outcomes. Am J Phys Med Rehabil. 2015 Feb;94(2):85-96; quiz 97-100. doi: 10.1097/PHM.0000000000000226. PMID 25569470
- [Result] Chan L, Sandel ME, Jette AM, Appelman J, Brandt DE, Cheng P, Teselle M, Delmonico R, Terdiman JF, Rasch EK. Does postacute care site matter? A longitudinal study assessing functional recovery after a stroke. Arch Phys Med Rehabil. 2013 Apr;94(4):622-9. doi: 10.1016/j.apmr.2012.09.033. Epub 2012 Nov 1. PMID 23124133
- [Result] Miller EL, Murray L, Richards L, Zorowitz RD, Bakas T, Clark P, Billinger SA; American Heart Association Council on Cardiovascular Nursing and the Stroke Council. Comprehensive overview of nursing and interdisciplinary rehabilitation care of the stroke patient: a scientific statement from the American Heart Association. Stroke. 2010 Oct;41(10):2402-48. doi: 10.1161/STR.0b013e3181e7512b. Epub 2010 Sep 2. No abstract available. PMID 20813995
- [Result] Winstein CJ, Stein J, Arena R, Bates B, Cherney LR, Cramer SC, Deruyter F, Eng JJ, Fisher B, Harvey RL, Lang CE, MacKay-Lyons M, Ottenbacher KJ, Pugh S, Reeves MJ, Richards LG, Stiers W, Zorowitz RD; American Heart Association Stroke Council, Council on Cardiovascular and Stroke Nursing, Council on Clinical Cardiology, and Council on Quality of Care and Outcomes Research. Guidelines for Adult Stroke Rehabilitation and Recovery: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2016 Jun;47(6):e98-e169. doi: 10.1161/STR.0000000000000098. Epub 2016 May 4. PMID 27145936
- [Result] MacDonald SL, Linkewich E, Bayley M, Jeong IJ, Fang J, Fleet JL. The association between inpatient rehabilitation intensity and outcomes after stroke in Ontario, Canada. Int J Stroke. 2024 Apr;19(4):431-441. doi: 10.1177/17474930231215005. Epub 2023 Dec 11. PMID 38078378
- [Result] Donkor ES. Stroke in the 21st Century: A Snapshot of the Burden, Epidemiology, and Quality of Life. Stroke Res Treat. 2018 Nov 27;2018:3238165. doi: 10.1155/2018/3238165. eCollection 2018. PMID 30598741
- [Result] Feigin VL, Brainin M, Norrving B, Martins S, Sacco RL, Hacke W, Fisher M, Pandian J, Lindsay P. World Stroke Organization (WSO): Global Stroke Fact Sheet 2022. Int J Stroke. 2022 Jan;17(1):18-29. doi: 10.1177/17474930211065917. PMID 34986727